CLINICAL TRIAL: NCT05481333
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of REGN7999, a TMPRSS6 Antagonist, in Healthy Adult Subjects
Brief Title: A Trial to Learn if REGN7999 is Safe and Well Tolerated, and How it Works in the Body of Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R7999-HV-2154; 2022-500398-15-00 (Other: EUCT Number)
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Non-menstruating; Transmembrane protease, serine 6 (TMPRSS6) antagonist; First in Human (FIH); Human monoclonal antibody (mAb)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- IV Cohort 1 (Experimental): Single dose REGN7999 or Placebo; randomized 3:1
  Interventions: Drug: REGN7999; Drug: Placebo
- IV Cohort 2 (Experimental): Single dose REGN7999 or Placebo; randomized 3:1
  Interventions: Drug: REGN7999; Drug: Placebo
- IV Cohort 3 (Experimental): Single dose REGN7999 or Placebo; randomized 3:1
  Interventions: Drug: REGN7999; Drug: Placebo
- IV Cohort 4 (Experimental): Single dose REGN7999 or Placebo; randomized 3:1
  Interventions: Drug: REGN7999; Drug: Placebo
- IV Cohort 5 (Experimental): Single dose REGN7999 or Placebo; randomized 3:1
  Interventions: Drug: REGN7999; Drug: Placebo
- SC Cohort 1 (Experimental): Single dose REGN7999 or Placebo; randomized 3:1
  Interventions: Drug: REGN7999; Drug: Placebo
- SC Cohort 2 (Experimental): Single dose REGN7999 or Placebo; randomized 3:1
  Interventions: Drug: REGN7999; Drug: Placebo
- SC Cohort 3 (Experimental): Single dose REGN7999 or Placebo; randomized 3:1
  Interventions: Drug: REGN7999; Drug: Placebo

INTERVENTIONS:
Drug: REGN7999 — Ascending IV or SC dose administered per protocol
Drug: Placebo — Ascending IV or SC dose administered per protocol

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single ascending intravenous (IV) and subcutaneous (SC) doses of REGN7999 in healthy adult participants.

The secondary objectives of the study are:

* To characterize the drug concentration profile of single doses of IV or SC REGN7999
* To assess the immunogenicity of single ascending SC or IV doses of REGN7999

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a body mass index between 18 and 32 kg/m2, inclusive
2. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and electrocardiogram (ECG)s performed at screening and/or prior to administration of initial dose of study drug
3. Is in good health based on laboratory safety testing obtained at the screening and baseline visits per the protocol
4. Hemoglobin, serum iron, transferrin, serum ferritin, and transferrin saturation, equal to or above the lower limit of the reference range for the participant's age and sex at the local labs, at screening, repeatable once during screening period
5. White blood cell (WBC) count, platelet count, red blood cell (RBC) count, hematocrit, and RBC hemoglobin not clinically significantly outside of the reference range in the judgment of the investigator at screening and baseline visits

Key Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Consistent with Clinical Trial Facilitation Group (CTFG) guidance, women of childbearing potential (WOCBP) who are unwilling to practice highly effective contraception, during the study through the end of study (EOS) visit. Highly effective contraceptive measures include:

   1. stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening;
   2. intra-uterine device (IUD); intra-uterine hormone-releasing system;
   3. bilateral tubal ligation or tubal occlusion;
   4. vasectomized partner (provided that the male vasectomized partner is the sole sexual partner of the WOCBP study participant and that the vasectomized partner has obtained medical assessment of surgical success for the procedure); and/or
   5. sexual abstinence as described in the protocol
3. In addition, premenopausal women whose method(s) of birth control is/are associated with ongoing menstruation (eg, combined hormonal contraceptive regimens associated with withdrawal bleeding, non-hormone-releasing IUD, bilateral tubal ligation, bilateral salpingectomy, vasectomized partner, sexual abstinence). Female participants must not be menstruating during the trial, due to being postmenopausal or due to permanent sterilization via hysterectomy, and/or bilateral oophorectomy, or amenorrheic due to use of hormone-releasing IUD, implantable device, or intake of continuous hormonal contraception
4. Sexually active male participants with WOCBP partners who are unwilling to use the following forms of medically acceptable birth control during the study through the EOS visit: vasectomy with medical assessment of surgical success OR consistent use of a condom
5. History of clinically significant cardiovascular (including congestive heart failure and angina), respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, infectious, autoimmune, oncologic, psychiatric or neurological disease, as assessed by the investigator, that may confound the results of the study or poses an additional risk to the participant by study participation.
6. History of chronic anemia, at any time in the past
7. History of RBC transfusion reaction
8. Whole blood donation within the previous 56 days or plasma donation within the previous 7 days prior to screening. Planning on whole blood or plasma donation at any time point during the study.
9. Has a history of significant multiple and/or severe allergies (eg, latex gloves), or has had an anaphylactic reaction to prescription or nonprescription drugs or food

Note: Other protocol-defined Inclusion and Exclusion Criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAEs) in participants treated with REGN7999 or placebo | Through the end of study visit, week 20
  IV cohorts 1 to 4 SC cohorts 1 and 2
Incidence and severity of TEAEs in participants treated with REGN7999 or placebo | Through the end of study visit, week 26
  IV cohort 5 and SC cohort 3

SECONDARY OUTCOMES:
Concentrations of REGN7999 in serum | Through the end of study visit, week 20
  IV cohorts 1 to 4 for SC cohorts 1 and 2
Concentrations of REGN7999 in serum | Through the end of study visit, week 26
  IV cohort 5 and SC cohort 3
Incidences of anti-drug antibodies (ADA) to REGN7999 over time | Through the end of study visit, week 20
  IV cohorts 1 to 4 for SC cohorts 1 and 2
Incidences of anti-drug antibodies (ADA) to REGN7999 over time | Through the end of study visit, week 26
  IV cohort 5 and SC cohort 3

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Drug Research Unit Gent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/